CLINICAL TRIAL: NCT07378267
Title: Effect of Intermittent Fasting and Mediterranean Diet on Body Composition and Nutritional Intake in Overweight and Obese Individuals: Randomized Trial
Brief Title: Effect of Intermittent Fasting and Mediterranean Diet on Body Composition and Nutritional Intake
Acronym: Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, SUHİDE BİLGE HORZUM, dietician, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023/54
Record Dates: First submitted 2026-01-17; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
Keywords: intermittent fasting; Mediterranean diet
MeSH Terms: conditions — Obesity; Overweight; Intermittent Fasting | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized trial using a dietary intervention method (Mediterranean Diet intervention group and Intermittent Fasting Diet group).
  First, inclusion criteria for randomization were determined, and 100 participants meeting these criteria who applied to a private diet clinic after a health screening from a family physician in Selçuklu district of Konya province will be assigned numbers. Individuals will be placed in the group corresponding to the dietary intervention group with the number they received in randomization. Dietary intervention will be applied to both groups in the study. After obtaining informed consent from the participants, an 8-week follow-up period will begin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet group (Active Comparator): Mediterranean diet
  Interventions: Other: Mediterranean diet
- intermittent fasting group (Active Comparator): intermittent fasting
  Interventions: Other: intermittent fasting

INTERVENTIONS:
Other: Mediterranean diet — The participants in the study were divided into two different diet groups: Mediterranean diet (MD) and intermittent fasting (IF). The "Harris Benedict" formula was used to calculate the Basal Metabolic Rate (BMR) of the individuals. For men, the BMR was calculated as 66.5 + (13.7516 × weight in kg) + (5.0033 × height in cm) - (6.755 × age in years); for women, the BMR was calculated as 655.1 + (9.5634 × weight in kg) + (1.8496 × height in cm) - (4.6756 × age in years). Physical activity level (PAL) was determined as follows: sedentary physical activity level 1-1.39; light physical activity level 1.4-1.59; moderate physical activity level 1.6-1.89; and heavy physical activity level 1.9-2.5. Total energy expenditure (TED) was calculated using the formula: TED (kcal/day) = BMR (kcal/day) x PAL (Ministry of Health, 2017). For the group following the Mediterranean diet, diet plans were prepared containing 35-40% carbohydrates, 15-20% protein, and 35-45% fat of daily energy. A nutritional pr
  Arms: Mediterranean diet group
Other: intermittent fasting — The participants in the study were divided into two different diet groups: Mediterranean diet (MD) and intermittent fasting (IF). The "Harris Benedict" formula was used to calculate the Basal Metabolic Rate (BMR) of the individuals. For men, the BMR was calculated as 66.5 + (13.7516 × weight in kg) + (5.0033 × height in cm) - (6.755 × age in years); for women, the BMR was calculated as 655.1 + (9.5634 × weight in kg) + (1.8496 × height in cm) - (4.6756 × age in years). Physical activity level (PAL) was determined as follows: sedentary physical activity level 1-1.39; light physical activity level 1.4-1.59; moderate physical activity level 1.6-1.89; and heavy physical activity level 1.9-2.5. Total energy expenditure (TED) was calculated using the formula: TED (kcal/day) = BMR (kcal/day) x PAL (Ministry of Health, 2017). Individuals in the intermittent fasting group also had time restrictions applied in addition to the Mediterranean diet group. Time preferences were determined as 16/8, 14
  Arms: intermittent fasting group

SUMMARY:
Cardiovascular diseases (CVD), cancer, diabetes, stroke, and chronic lung diseases are non-communicable diseases (NCDs) and account for a significant portion of deaths worldwide. In Turkey, it is estimated that 90% of all deaths are due to NCDs, with 34% due to CVD, 23% due to cancer, 7% due to chronic lung disease, and 5% due to diabetes.

Inadequate and unbalanced nutrition and lack of physical activity contribute to the development of non-communicable diseases. Risk factors such as hypertension, hypercholesterolemia, and obesity are effective in increasing NCDs. In Turkey, it has been found that 32% of NCD-related deaths in individuals over 18 years of age and 10% in adolescents aged 10-19 years are due to obesity risk factors.

All overweight and obese adults with a Body Mass Index (BMI) ≥25 are at risk of developing hypertension, hypercholesterolemia, type 2 diabetes, and CVD. Preventing obesity is effective in preventing these diseases. Weight loss is important in the treatment and prevention of obesity. Changes in body weight are focused on changes in diet and physical activity. Creating an energy deficit is necessary to achieve weight loss, and there are different dietary approaches to reduce energy intake. The Mediterranean diet model and the Intermittent Fasting model are important and being researched in this context.

DETAILED DESCRIPTION:
The Mediterranean diet, based on the nutritional patterns of people living in the Mediterranean region, has been found to have a different dietary style and may be effective against CHD and many other diseases. The Mediterranean diet is a model based on a high ratio of monounsaturated and saturated fats, high consumption of legumes, high consumption of fruits and vegetables, low consumption of meat and meat products, and moderate consumption of milk and dairy products. It is thought that the Mediterranean diet can be effective both in preventing diseases and in managing the disease process. In addition, the Mediterranean diet has been used in calorie-restricted diet models due to its effect on obesity and body composition. When the studies in the literature are examined; in a meta-analysis, weight loss was observed in Mediterranean diet models with energy restriction. In an intervention study based on the Mediterranean diet model in obese patients with metabolic syndrome, significant changes occurred in BMI, total fat percentage, total lean mass percentage, and abdominal fat percentage. Another study showed statistically significant changes in body weight and BMI in individuals who underwent Mediterranean diet intervention. Along with this change in body weight, the group with more than 5% weight loss showed a decrease in total cholesterol and triglyceride levels and values such as HOMA-IR in blood parameters. Furthermore, another meta-analysis found that some studies showed that the Mediterranean diet significantly reduced the likelihood of overweight/obesity, supported weight loss, or caused greater weight loss than the control diet, while other studies found no significant association between the Mediterranean diet and overweight/obesity.

Fasting is known as one of the oldest traditions in the world and is practiced among various communities for cultural or religious reasons. Fasting has also been used in the past as a method of treating illnesses. Hippocrates, considered the father of modern medicine, emphasized the importance of fasting during illness with his statement, "To eat when you are sick is to feed your illness". Intermittent fasting, that is, periods of voluntary abstinence from food and drink, is an ancient practice followed in different forms by many populations worldwide. Intermittent fasting involves fasting or restricted eating at certain times of the day or on certain days of the week. Alternate-day fasting involves alternating days when food and drinks are consumed with days when energy-containing foods or drinks are not consumed. In alternate-day fasting, approximately 20-25% of energy requirements are met on fasting days. Modified fasting is also known as the 5:2 method. This dietary model involves a very low-calorie diet on 2 non-consecutive days of the week, and normal energy requirements without energy restriction on the other 5 days. Another approach is time-restricted eating, which is used to describe an eating pattern where food intake is limited to a time window of 8 hours or less each da. Welton et al. reported that the ideal fasting period for positive weight change is 16 hours. In recent years, small-scale human studies demonstrating the importance of time-ricted eating have become widespread. Most of these studies, as in animal studies, have revealed the beneficial aspects of intermittent fasting in human metabolism. With time-restricted eating, reductions in energy intake, body weight, body fat, blood sugar, triglycerides, glucose tolerance, and inflammatory markers have been observed. Among fasting methods are religious fasts, such as Ramadan, which allow eating after sunset and before dawn. Since the fasting and eating periods last approximately 12 hours and the amount of energy given is not limited, it is a type of time-restricted eating.

Intermittent fasting, which has become a popular topic recently, is an alternative energy restriction method. Time-restricted eating, alternate-day fasting, the 5:2 diet, and Ramadan fasting are the most frequently used fasting protocols in the literature. Although daily energy restriction is the most commonly used diet model for achieving weight loss and improving body composition and metabolic health, intermittent fasting practices have become a focus of interest in recent years.

A review of studies in the literature revealed statistically significant differences in pre- and post-intervention body weight and BMI in 33 adults who underwent an 8-hour time-restricted feeding model for four weeks. A randomized controlled trial of 16 men and women (BMI 20-39 kg/m²) conducted over 10 weeks examined changes in body composition between the intervention and control groups using a time-restricted feeding model without energy restriction. According to Liu et al., no significant differences were found between the experimental and control groups in terms of reduction in body weight, body fat, or metabolic risk factors in obese individuals who underwent a time-restricted feeding model. A significant decrease in body fat percentage was observed in the time-restricted feeding model compared to the control group, while there was no significant change in body weight in either group. In another study, 101 overweight and obese adults were randomized into an alternate-day fasting group (n=34), a 16/8 time-restricted feeding group (n=33), and a control group (n=34). In the alternating-day fasting and 16/8 time-restricted eating groups, reductions in body weight, body mass index, and waist circumference were found to be more significant compared to the control group. Furthermore, the reductions in body weight and BMI in the alternating-day fasting group were more significant than those in the 16/8 group. In another randomized controlled trial of 40 obese young people aged 18-25, the intervention group underwent a 5:2 intermittent fasting diet, while the control group continued their previous eating habits. After a four-week intervention, the group undergoing 5:2 intermittent fasting showed a statistically significant decrease in energy intake and BMI compared to the control group. In contrast, Witjaksono et al. monitored weight loss in 50 obese participants using a 5:2 modified diet model (n=25) and a control group (n=25). While there were no significant changes in fat mass, lean mass, skeletal muscle, and BMI between the groups, reductions in carbohydrate, protein, and fat intake were statistically significant in both groups.

In conclusion, the prevalence of noncommunicable diseases is increasing today, and obesity is among the important risk factors for these diseases. While many methods are used in the treatment of obesity, medical nutritional therapies are also important. Different methods are used in medical nutritional therapies for obesity, including calorie-restricted Mediterranean diets and time-restricted eating models, which are one of the intermittent fasting models. This study aimed to examine the effect of dietary models on body composition and dietary intake in the management of obesity.

ELIGIBILITY:
Inclusion Criteria:

Being between 18-65 years old

Having a BMI value between 27 kg/m2 - 35 kg/m2

HBA1C levels between 3.9-6.1

HOMA IR <2.5

Not having any conditions that impair reality testing and cognitive functions, preventing interviewing or completing scales

Being literate

Having signed the informed consent form by agreeing to participate in the research

Exclusion Criteria:

Being pregnant or breastfeeding,

Liver and kidney disease,

Use of insulin and oral antidiabetic drugs,

Defined as a psychiatric illness diagnosed by a physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Adult Nutrition Knowledge Level (ADHL) Scale | 8 weeks
  The survey form containing Basic Nutrition and Food-Health Information will be completed. Participants who marked "Strongly Agree" for correct statements received 4 points, those who marked "Agree" received 3 points, those who marked "Neither Agree nor Disagree" received 2 points, those who chose "Disagree" received 1 point, and those who chose "Strongly Disagree" received 0 points. Items 1, 3, 6, 8, 13, 16, 19, and 20 of the scale are reverse scored. The highest possible score for the basic nutrition section is 80; the highest possible score for the food preference section is 48. A basic nutrition score of <45 is considered poor, 45-55 is considered average, 56-65 is considered good, and 65 and above is considered very good. In terms of food preference scores, a score of <30 is considered poor, 30-36 points are considered average, 37-42 points are considered good, and 42 points and above are considered very good.
Body fat percentage (%Fat) | 8 weeks
  Individuals' body weights and body compositions will be measured using foot-to-foot bioelectrical impedance analysis (BIA).
  Body fat percentage (%Fat) will be measured using TANITA MC 580.

SECONDARY OUTCOMES:
Body fat mass (kg) | 8 weeks
  Individuals' body weights and body compositions will be measured using foot-to-foot bioelectrical impedance analysis (BIA).
  Body fat mass (kg) will be measured using TANITA MC 580.
Weight | 8 weeks
  Individuals' body weights and body compositions will be measured using foot-to-foot bioelectrical impedance analysis (BIA).
  Weight will be measured using TANITA MC 580.
Body mass index (BMI) | 8 weeks
  Body mass index (BMI) will be calculated using the equation where body weight is divided by the square of height in meters, and will be evaluated according to the World Health Organization's classification for adults.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Bayrak, assistant professor, Study Director — Selcuk University
Locations (1):
- Eda Ocak Nutrition and Diet Consultancy, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication.
Supporting Information: Study Protocol, ICF
Time Frame: February 2023 - November 2023
Access Criteria: Access criteria will be shared with researchers who meet the following conditions:
  Being employed by a recognized academic institution, university, research hospital, or public research organization; Providing documentation that the study in which the requested data will be used has scientific, ethical, and social benefit purposes; Submitting a research protocol approved by the relevant institution or ethics committee; Committing that the data will be used only for secondary analysis or meta-analysis.

REFERENCES:
- [Result] Antoni, R., Robertson, T. M., Robertson, M. D., Johnston, J. (2018). A pilot feasibility study exploring the effects of a moderate time-restricted feeding intervention on energy intake, adiposity and metabolic physiology in free-living human subjects. 7. doi:https://doi.org/10.1017/jns.2018.13